CLINICAL TRIAL: NCT04754425
Title: A Study of Erdafitinib in Castration-Resistant Prostate Cancer Patients Evaluating Markers of Bone Remodeling and FGF Signaling in Plasma and Bone Marrow
Brief Title: Erdafitinib for the Treatment of Patients With Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0953; NCI-2021-00663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0953 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Castration-Resistant Prostate Carcinoma; Castration-Resistant Prostate Carcinoma Refractory to Second-Generation Androgen Receptor Axis-Targeted Agents; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Adenocarcinoma; Metastatic Prostate Small Cell Neuroendocrine Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (erdafitinib, biospecimen collection) (Experimental): Patients receive erdafitinib PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may also undergo collection of blood and bone marrow via biopsy and aspirates.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Erdafitinib

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and bone marrow
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ-42756493

SUMMARY:
This phase II trial studies the effect of erdafitinib in treating patients with prostate cancer that grows and continues to spread despite the surgical removal of the testes or drugs to block androgen production (castration-resistant). Erdafitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving erdafitinib may help control disease in patients with castration-resistant prostate cancer. In addition, studying samples of blood, tissue, plasma, and bone marrow from patients with castration-resistant prostate cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate efficacy of erdafitinib in subjects with advanced prostate cancer who have progressed on a second-generation androgen receptor (AR)-targeting agents (SART).

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate II. To measure Time on Treatment (ToT) as a surrogate of clinical efficacy and Progression-Free Survival (PFS) III. To measure PFS. IV. To correlate bone specific alkaline phosphatase (BAP) modulation with response, ToT and PFS.

V. To correlate prostate specific antigen (PSA) modulation with response, ToT and PFS.

VI. To characterize the safety profile of subjects treated with erdafitinib. VII. To measure overall survival. VIII. To collect and archive bone marrow biopsies and aspirates, serum and plasma in study patients for later hypothesis generating associations.

EXPLORATORY OBJECTIVE:

I. To evaluate DNA, ribonucleic acid (RNA), or protein biomarkers in tissue and blood samples which potentially predict tumor response or resistance to erdafitinib.

OUTLINE:

Patients receive erdafitinib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may also undergo collection of blood and bone marrow via biopsy and aspirates.

After completion of study treatment, patients are followed up at 30 days, every 16 weeks for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically proven adenocarcinoma or small cell of the prostate with evidence for skeletal metastases on bone scan and/or computed tomography (CT)/positron emission tomography (PET)/magnetic resonance imaging (MRI) scan. Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Serum testosterone levels =< 50 ng/ml and maintenance of castration with luteinizing hormone-releasing hormone (LHRH) agonist/antagonist or orchiectomy
* Patients must have documented evidence of progressive disease as defined by any of the following:

  * PSA progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least >= 1.0 ng/mL
  * New or increasing non-bone disease (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria)
  * Positive bone scan with 2 or more new lesions (Prostate Cancer Working Group 3 [PCWG3])
* Prior treatment with a second-generation AR-targeting agent (e.g. abiraterone acetate, enzalutamide, apalutamide) is required. Patients may have received up to two such agents
* Patients may have received prior treatment with immunotherapies (sipuleucel-T, checkpoint immunotherapies) or bone targeting therapies (radium-223)
* Both chemotherapy-naive and patients previously treated with chemotherapy are eligible. Chemotherapy pretreated patients may have received a maximum of two prior systemic cytotoxic chemotherapies completed at least 3 weeks prior to initiation of study treatment
* Hemoglobin >= 8.0 g/dL
* Platelet count >= 75,000/uL
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Calculated creatinine clearance (Cockcroft-Gault Equation) >= 40 mL/min
* Serum potassium >= institutional lower limit of normal (ILLN)
* Serum magnesium >= ILLN
* Serum albumin >= 3.0 g/dL
* Serum bilirubin < 1.5 x institutional upper limit of normal (IULN) (except for patients with known Gilbert's disease)
* Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x IULN for patients without liver metastases. For patients with liver metastases AST or ALT < 5 x IULN is allowed
* Able to swallow study drugs whole as a tablet/capsule
* Patients must agree to tissue and blood collection for correlative studies at the specified time points
* Male subject with a female partner of childbearing potential or pregnant must agree to use two acceptable methods of contraception and not to donate sperm from time of screening until 3 months after the last dose of study treatments

Exclusion Criteria:

* Radiation therapy to primary tumor or metastatic sites within 2 weeks of cycle 1, day 1
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 30 days prior to randomization
* A malignancy (other than the one treated in this study) which required radiotherapy or systemic treatment within the past 1 year, or has a >= 30% probability of recurrence within 24 months (except for non-melanoma skin cancer or Ta urothelial carcinomas)
* Chronically uncontrolled hypertension, defined conventionally as consistent systolic pressures above 160 or diastolic pressures above 100 despite anti-hypertensive therapy. Note that this is NOT a criterion related to particular blood pressure (BP) results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes. (For example doctor's visit related stress i.e. "white coat syndrome")
* Eye conditions likely to increase the risk of eye toxicity including

  * Corneal or retinal abnormality likely to increase the risk of eye toxicity, or lens conditions such as: untreated mature or hypermature senile cataract, affecting visual acuity that impair the ability to interpret the Amsler grid test
  * History of central serous retinopathy (CSR) or retinal vascular occlusion (RVO)
  * Active wet, age-related macular degeneration (AMD)
  * Diabetic retinopathy with macular edema (non-proliferative)
  * Uncontrolled glaucoma (per local standard of care)
  * Corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events
* History of uncontrolled cardiovascular disease including:

  * Unstable angina, myocardial infarction, ventricular fibrillation, Torsades de Pointes, cardiac arrest, or known congestive heart failure class III-V within the preceding 3 months; cerebrovascular accident or transient ischemic attack within the preceding 3 months
  * Mobitz II second degree heart block or third degree heart block
  * Corrected QT interval (QTc) prolongation as confirmed by triplicate assessment at screening (Fridericia; QTc > 480 milliseconds)
  * Pulmonary embolism or other venous thromboembolism (VTE) within the preceding 2 months
* Known active autoimmune deficiency syndrome (AIDS) (human immunodeficiency virus [HIV] infection), unless the subject has been on a stable anti-retroviral therapy regimen for the last 6 months or more, has had no opportunistic infections in the last 6 months, and has CD4 count > 350
* Known active hepatitis B or C infection (subjects with history of hepatitis C infection but negative hepatitis C virus polymerase chain reaction ([PCR] test and subjects with hepatitis B with positive hepatitis B surface antibody are allowed)
* Not recovered from reversible toxicity of prior anticancer therapy (except toxicities which are not clinically significant such as alopecia, skin discoloration, grade 1 neuropathy, grade 1-2 hearing loss)
* Impaired wound healing capacity defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or unhealed incisions
* Major surgery within 4 weeks before randomization
* Untreated symptomatic spinal cord compression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Bone specific alkaline phosphatase (BAP) modulation | Up to 5 years
  Will assess modulation of BAP under the influence of treatment. Calculated as the maximal percentage change (decrease versus increase) on treatment. BAP in blood samples will be used for the primary analysis. Proportion of patients with BAP reduction along with the 95% confidence interval (95% CI) will be estimated.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  Defined as (a) the proportion of subjects with soft tissue disease who achieve complete response or partial response, as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 by the investigator and (b) the proportion of subjects with improvement in bone imaging as assessed by the principal investigator. Will be estimated with proportion and its corresponding 95% CI.
Time on treatment | Duration in weeks/months from the time of treatment start until the patient goes off treatment for any reason, assessed up to 5 years
  Measured as a surrogate of clinical efficacy and progression-free survival (PFS). Will be estimated using the method of Kaplan and Meier and the effects of potential.
Progression-free survival | Duration in weeks/months from the time of treatment start to the date of disease progression or death, whichever is reported first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier and the effects of potential.
Prostate specific antigen modulation | Up to 5 years
  Calculated as the maximal percentage change (decrease versus increase) on treatment.
Incidence of adverse events | Up to 5 years
  Will be reported by their National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 term by grade and attribution.
Overall survival | Duration in weeks/months from the time of treatment start to the date of death, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier and the effects of potential.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT04754425/ICF_000.pdf